CLINICAL TRIAL: NCT06536010
Title: Clinical Trial Protocol for the Combined Use of Azacitidine, Venetoclax, and Granulocyte Colony-Stimulating Factor in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML) (Phase IIb, Single-arm, Prospective, Single-center Study)
Brief Title: Clinical Trial Protocol for the Combined Use of VAG in the Treatment of ND-AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Xiaotian (Other)
Responsible Party: Sponsor-Investigator, Yang Xiaotian, Principal Investigator, The Second People's Hospital of Huai'an
Organization: The Second People's Hospital of Huai'an (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEYLL202403
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VAG regimen in the treatment of newly diagnosed acute myeloid leukemia (AML) (Experimental): AZA: 75mg/m2 on days 1-7 VEN: 100mg on day 1, 200mg on day 2, 400mg on days 3-28 G-CSF: 50-600ug/day, starting on day 1 (adjusted based on WBC count of 10-25*10E9/L)
  In the induction phase of the ND-AML treatment protocol, VEN+AZA+G-CSF is administered. At the end of the induction phase, the efficacy is evaluated. If the patient achieves complete remission (CR), the original treatment protocol is continued for consolidation. If the patient achieves partial remission (PR), the original treatment protocol is repeated for induction until the patient achieves CR or shows no response (NR), progressive disease (PD), or relapse (PR/NR/PD). If the patient shows no response or progressive disease, the study is concluded.
  Interventions: Drug: Venetoclax 100 mg d1，200 mg d2，400 mg d3-28；

INTERVENTIONS:
Drug: Venetoclax 100 mg d1，200 mg d2，400 mg d3-28； — VAG in the induction phase of the ND-AML treatment protocol
  Other Names: AZA 75mg/m2 on days 1-7; G-CSF: 50-600ug/day, starting on day 1 (adjusted based on WBC count of 10-25*10E9/L)

SUMMARY:
This is a clinical efficacy study evaluating the VAG regimen in the treatment of newly diagnosed acute myeloid leukemia (AML).

The main objectives of the study are to assess the efficacy and safety of the VAG regimen and to explore the synergistic mechanisms of VAG in combating AML.

DETAILED DESCRIPTION:
This study is a single-arm, prospective, single-center phase IIb clinical efficacy study evaluating the therapeutic effects of azacitidine and venetoclax in combination with granulocyte colony-stimulating factor for the treatment of newly diagnosed acute myeloid leukemia (AML).

Acute myeloid leukemia (AML) is a malignant disease originating from myeloid hematopoietic stem/progenitor cells. It is highly aggressive, and patients have a very low survival rate. The 5-year survival rate for diagnosed AML patients is approximately 29%, with only 5-15% for patients aged 60 and above. Currently, the 3+7 regimen is the first-line induction chemotherapy for newly diagnosed AML patients, with about 60-80% of young patients (<60 years old) and 40-60% of elderly patients (≥60 years old) achieving complete remission (CR). However, among AML patients receiving the 3+7 regimen, those with poor physical condition or high-risk cytogenetics have a worse prognosis. Therefore, there is a need to explore new treatment regimens that are less intensive but still effective.

Venetoclax is an oral selective Bcl-2 inhibitor. Multiple studies and clinical trials have demonstrated that Venetoclax, in combination with demethylating agents or low-dose cytarabine (LDAC), has synergistic anti-tumor effects and achieves higher treatment response and disease-free survival rates in AML patients. The results of the VIALE-A study showed that the median overall survival (OS) time with Venetoclax plus Azacitidine (AZA) was 14.7 months compared to 9.6 months with Azacitidine alone (P<0.001). The median duration of remission was 17.5 months with Venetoclax plus Azacitidine compared to 13.4 months with Azacitidine alone, and the CR+CRi rates were 66.4% and 28.3%, respectively (P<0.001). This combination significantly improves the overall survival of AML patients, with high response rates and good safety profile. In October 2020, the U.S. Food and Drug Administration approved the use of Venetoclax in combination with Azacitidine, Decitabine, or LDAC for the treatment of newly diagnosed AML patients aged 75 years or older or those who are unfit for intensive induction chemotherapy due to comorbidities. The Venetoclax plus Azacitidine regimen was also included in the AML NCCN guidelines in 2020. However, while Venetoclax in combination with demethylating agents is recommended for the treatment of elderly AML patients, there is currently a lack of research data for its use in young AML patients. The results of a phase II clinical trial presented at the 2022 ASH Annual Meeting, evaluating Venetoclax plus hypomethylating agents in young adults with newly diagnosed AML and adverse ELN risk, showed a complete remission with incomplete hematologic recovery (CRc) rate of 78% after one cycle of treatment, with a minimal residual disease (MRD) negativity rate of 77%. After two cycles of treatment, the CRc rate was 91.9% with an MRD negativity rate of 82.3%. The CRc rates for favorable, intermediate, and adverse risk groups were 69.6%, 75.4%, and 61.3%, respectively. Although the combination of Venetoclax and demethylating agents has shown promising efficacy, there are still limitations such as adverse events including thrombocytopenia (46%), nausea (44%), constipation (43%), neutropenia (42%), febrile neutropenia (42%), diarrhea (41%), and tumor lysis syndrome (TLS), as well as suboptimal achievement of MRD negativity and depth of remission after induction therapy.

Granulocyte colony-stimulating factor (G-CSF) is expressed by almost all AML cells and binds to its receptor, G-CSFR. In pre-activation regimens, G-CSF induces tumor cells in the quiescent phase (G0/G1) to enter the proliferative phase (S phase), enhancing the cytotoxic effect of chemotherapy drugs on tumor cells, improving the efficacy of chemotherapy, and reducing adverse reactions. A study conducted by Tang Xiaowen's team at the First Affiliated Hospital of Soochow University on the efficacy and safety of decitabine (DAC) combined with HAAG in the treatment of newly diagnosed acute myeloid leukemia showed that after one cycle of DAC+HAAG induction therapy in 50 patients, 48 patients (96%) achieved complete remission (CR)/CR with incomplete blood count recovery (CRp)/CR with incomplete count recovery and incomplete marrow recovery (CRi), and 2 patients (4%) achieved partial remission (PR). The median time to recovery of white blood cell count, platelet count, and hemoglobin was 17.5 days, 19.0 days, and 20.0 days, respectively. Only 16% (8/50) and 6% (3/50) of patients experienced grade 3-4 infections and bleeding, while non-hematologic toxicities were mainly grade 1-2 and resolved after symptomatic treatment.

The combination of venetoclax and hypomethylating agents is the most common approach, which synergistically induces cell apoptosis and reduces MCL-1 levels, thereby overcoming resistance to BCL-2 inhibitors. Additionally, the combination interferes with the energy metabolism of leukemia cells and targets leukemia stem cells. However, there is currently no research on the combination of azacitidine, venetoclax, and G-CSF. The investigators has conducted a preliminary clinical study on the VAG regimen (azacitidine, venetoclax, and granulocyte colony-stimulating factor) for newly diagnosed AML, which has shown promising results. We plan to expand the sample size and further investigate its mechanism of tumor cell killing.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, regardless of gender.
* Diagnosis of AML (excluding APL) according to the 2022 World Health Organization (WHO) diagnostic criteria.
* ECOG performance status of 0-2.
* For female participants of childbearing potential or male participants with female partners of childbearing potential, effective contraceptive measures must be taken throughout the entire treatment period and for 6 months after the treatment period.
* Expected survival of at least 3 months.
* Ability to understand and willingness to participate in the study, and signing an informed consent form.

Exclusion Criteria:

* Acute promyelocytic leukemia (M3 subtype).
* Central nervous system leukemia.
* Severe uncontrolled infection or other major diseases.
* Heart failure: Ejection fraction (EF) < 50%, New York Heart Association (NYHA) class II or above.
* Impaired liver or kidney function: Serum total bilirubin ≥ 2.0 mg/dl, AST ≥ 3 times the upper limit of normal, serum creatinine clearance rate (Ccr) ≥ 50 ml/min, arterial oxygen saturation (SpO2) < 92%.
* Human immunodeficiency virus (HIV) positive.
* Active hepatitis B or C.
* Pregnant or lactating women.
* Other conditions in which the investigator deems the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) | The period of 2 months from the start of treatment.
  A. No symptoms or signs of leukemia cell infiltration, normal or near-normal life; B. Blood counts: Hb ≥ 100g/L (males) or ≥ 90g/L (females and children), absolute neutrophil count ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L. No leukemia cells in peripheral blood leukocyte classification; C. Bone marrow morphology: Less than or equal to 5% of myeloblasts (type I + type II) (primitive monocytes + immature monocytes or primitive lymphocytes + immature lymphocytes), normal red blood cells and megakaryocytes; D. No extramedullary leukemia (no lymphadenopathy, splenomegaly, skin/gum infiltration, testicular masses, central nervous system involvement).

SECONDARY OUTCOMES:
Partial Remission (PR) | The period of 1 month from the start of treatment.
  Myeloblasts (type I + type II) (primitive monocytes + immature monocytes or primitive lymphocytes + immature lymphocytes) > 5% but ≤ 20%; or one of the following criteria is met in clinical, blood counts, and bone marrow morphology for complete remission.
Complete Remission with incomplete blood count recovery (CRi) | The period of 1 month from the start of treatment.
  PLT < 100 × 109/L or NE < 1.5 × 109/L. Other criteria for CR should be met.
Overall Response Rate (ORR) | The period of 4 months from the start of treatment.
  CR+CRi+MLFS+PR
Morphologic leukemia-free state (MLFS) | The period of 1 month from the start of treatment.
  < 5% of primitive cells in bone marrow; no immature cells with Auer rods; no persistent extramedullary leukemia; no requirement for normal blood cell recovery.
Overall survival, OS | The period of 2 years from the start of treatment.
  The time from the start of treatment to death or the end of follow-up, evaluated at 2 years after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Huai'an Second People's Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided